CLINICAL TRIAL: NCT06672575
Title: A Phase I/II Study of IVONESCIMAB in Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1277; NCI-2024-09210 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Ivonescimab (Experimental): Participants will be enrolled in either Phase 1 or Phase 2 depending on when they join the study.
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — Participante will recived an infusion by vein

SUMMARY:
The goal of Phase 1 of this clinical research study is to find the highest tolerable dose and the recommended Phase 2 dose of ivonescimab that can be given to patients who have recurrent glioblastoma.

The goal of Phase 2 of this clinical research study is to learn if the recommended Phase 2 dose of ivonescimab found in Phase 1 can help to control the disease.

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the safety and tolerability of ivonescimab in adult patients with recurrent glioblastoma
* To determine the median progression free survival and progression free survival rate at 6 months of ivonescimab in adult patients with recurrent glioblastoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Karnofsky Performance Status (KPS) of 60 or greater
3. Recurrent supratentorial Glioblastoma that has progressed following standard therapy; patients must have previously been treated with radiation with or without temozolomide.

   1. Patients will be eligible at first or second recurrence.
   2. Patients must be greater than 12 weeks from completion of initial chemoradiation at the time of progression, with the exception that patients with biopsy-confirmed recurrent disease prior to this time window can be enrolled.
4. Diagnosis of Glioblastoma IDH-wildtype, WHO Grade 4 consistent with WHO CNS 2021 criteria. This will include patients with a diagnosis of molecular glioblastoma.
5. Measurable or evaluable disease per RANO criteria
6. A baseline MRI Brain no more than 14 days prior to study enrollment
7. Adequate Organ Function, with screening labs performed within 14 days of treatment initiation:

   a. Hematology (no blood transfusions or growth factor therapy used within 7 days of the screening CBC): i. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L ii. Platelet count ≥ 100 × 109/L iii. Hemoglobin ≥ 9.0 g/dL b. Kidneys: i. Creatinine clearance* (CrCL) ≥ 50 mL/min using the Cockcroft-Gault formula or estimated glomerular filtration rate (eGFR) value ≥50 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation (adjustment by BSA is not required for eGFR)

   CrCL or eGFR can be determined using the calculator from the National Kidney Foundation website (www.kidney.org).

   ii. Urine protein < 2+ or 24-hour urine protein quantification < 1.0 g or Urine protein/Creatinine ratio ≤ 1mg/mg (≤ 113.2mg/mmol) c. Liver: i. Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); For patients with confirmed/suspected Gilbert syndrome, TBIL ≤3 × ULN ii. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN d. Coagulation: prothrombin time (PT) or international normalized ratio (INR)
   * 1.5 × ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy or prophylactic coagulation)
8. Female patients of childbearing age must have negative serum pregnancy test results before randomization or per region-specific guidance documented in the informed consent and a negative urine pregnancy test on the day of first dose prior to dosing.
9. Female patient of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 120 days after the last dose of the ivonescimab.
10. Male patients of childbearing potential having sex with a female partner of childbearing potential must agree to use an effective method of contraception from the beginning of screening until Day 120 after the last dose of ivonescimab.
11. Ability to understand and willingness to sign informed consent form prior to the initiation of study and any study procedures.

    1. Participants with cognitive impairment may be enrolled. The formal consent for such participants will be obtained from their legally authorized representative. However, participants will be informed about the research to the maximum extent compatible with their understanding. Assent will be obtained from such participants who will sign and date the consent form if capable.
    2. Non-English speakers are allowed to enroll provided consent and all visits will be conducted with a medical interpreter.

Exclusion Criteria:

1. Major surgical procedures or serious trauma, or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator).

   Minor local procedures (excluding central venous catheterization and port implantation).
2. Currently pregnant or breastfeeding.
3. History of bleeding tendencies or coagulopathy and/or clinically significant bleeding symptoms, including but not limited to:

   a. Significant intracranial hemorrhage
   1. Note: Patients with clinically asymptomatic presence of hemosiderin, resolving postoperative changes or punctate intratumoral hemorrhage are permitted
   2. Gastrointestinal bleeding

   b. Hemoptysis (defined as coughing up ≥ 0.5 teaspoon of fresh blood or small blood clots) Note: transient hemoptysis associated with diagnostic bronchoscopy is allowed. c. Nasal bleeding /epistaxis (bloody nasal discharge is allowed) d. Need for therapeutic anticoagulant therapy Note: Prophylactic anticoagulation for DVT/PE or to maintain venous patency is allowed.
4. Current hypertension with systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
5. Is receiving dexamethasone >2mg daily, or the corticosteroid equivalent thereof.
6. History of major diseases, specifically:

   1. Unstable angina, myocardial infarction, congestive heart failure (New York Heart Association [NYHA] classification ≥ grade 2) or vascular disease (eg, aortic aneurysm at risk of rupture), or other cardiac impairment that may affect the safety evaluation of the study drug (eg, poorly controlled arrhythmias, myocardial ischemia)
   2. History of esophageal gastric varices, severe ulcers, wounds that do not heal, abdominal fistula, intra-abdominal abscesses, or acute gastrointestinal bleeding
   3. History of arterial thromboembolic event, venous thromboembolic event of Grade 3 and above as specified in National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy
   4. Acute exacerbation of chronic obstructive pulmonary disease within 4 weeks beforerandomization
   5. History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection)
7. History of other malignancy diagnosed or requiring treatment within the past 3 years prior to enrolment, with the exception of those with negligible expected risk of metastasis or death (including adequately treated non- melanoma skin cancer or cervical carcinoma in situ).
8. History of prior treatment of GB with anti-VEGF and/or anti-PD-1/PDL-1 agents, including monotherapy with either category or combinations thereof.
9. Has received prior interstitial brachytherapy, interstitial thermal therapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced deliver. Prior treatment with Gliadel ® wafers will be excluded. Concurrent use of devices such as Tumor Treating Fields is not permitted.
10. Has known leptomeningeal disease, gliomatosis cerebri, extracranial disease, or multicentric disease (regionally multifocal enhancing disease with continguous T2/FLAIR is permitted to be enrolled)
11. Uncontrolled seizures after best medical therapy or other neurological conditions including clinically significant autoimmune neurological disorders which can increase risk for adverse effects or confound assessment of study outcomes as determined by the treating physician and PI
12. History of clinically significant autoimmune disease including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, granulomatosis with polyangiitis, Sjogren's syndrome, GuillainBarré syndrome, multiple sclerosis, vasculitis or glomerulonephritis

    1. Patients with a history of autoimmune hypothyroidism may be eligible if on a stable dose of thyroid replacement hormone
    2. Patients with controlled Type 1 diabetes mellitus may be eligible if on a stable insulin regimen
    3. Patients with dermatologic disorders (e.g., eczema) may be eligible if well controlled at baseline and not requiring systemic treatment or other treatments beyond low potency topical steroids
13. Has contraindication for undergoing MRI scans or receiving MRI contrast.
14. History of stroke or TIA within 6 months prior to study enrolment.
15. Imaging during the screening period shows that the patient has:

    1. Radiologically documented evidence of major blood vessel invasion or encasement by cancer
    2. Radiographic evidence of intratumor cavitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Anuj D Patel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org